CLINICAL TRIAL: NCT00972218
Title: Efficacy of Adalimumab (Humira®) in Spondyloarthritis Related to Crohn's Disease
Brief Title: Effectiveness and Safety of Spondylitis Related to Inflammatory Bowel Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty with enrollment
Sponsor: University of Alberta (Other)
Collaborators: Abbott (Industry)
Responsible Party: Walter P. Maksymowych, University of Alberta
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A10-456
Record Dates: First submitted 2009-08-31; First posted 2009-09-04 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Spondyloarthritis; Crohn's Disease
Keywords: Spondyloarthritis; Ankylosing Spondylitis; Crohn's disease; adalimumab; treatment
MeSH Terms: conditions — Spondylarthritis; Crohn Disease; Spondylitis, Ankylosing | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enteropathic spondyloarthritis (Experimental): Patients have concomitant inflammatory spinal symptoms and inflammatory bowel disease.
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Adalimumab subcutaneous injections 40 mg dose every other week for 24 weeks
  Other Names: Humira

SUMMARY:
Adalimumab is an antibody treatment that targets and neutralizes a molecule produced in the body that is associated with inflammation, tumor necrosis factor (TNF). This molecule is an important factor in causing the inflammation seen in people with a form of inflammatory spinal arthritis called spondylitis as well as inflammation in the bowel called Crohn's disease. Spondylitis and Crohn's disease tend to go together and this study will assess to what degree this treatment is effective for those patients that have both disorders at the same time.

DETAILED DESCRIPTION:
The primary objective of the present study is to assess the efficacy of adalimumab in ameliorating the signs and symptoms of spondyloarthritis associated with CD. Although AS patients with IBD were recruited in phase III trials of anti-TNF therapy and shown to respond to treatment, this has not been established in a cohort of patients with exclusive enteropathic spondyloarthritis. Evaluation of such a cohort will address several important issues:

* Firstly, it will answer the question of whether or not patients with enteropathic spondyloarthritis respond to treatment with adalimumab.
* Secondly, since patients with IBD represent a cohort at high risk of developing spondyloarthritis, this approach will allow the study of the efficacy of adalimumab in patients with pre-radiographic inflammatory back pain as determined by clinical, laboratory, and radiological outcomes. In particular, the use of MRI as an outcome measure will be explored. In addition, this will allow the further evaluation of diagnostic criteria for pre-radiographic AS.
* Thirdly, the efficacy of adalimumab in treating IBD associated with SpA has not been previously determined. It has been assumed that the response should be the same as that observed in idiopathic disease. However, it is important to note that the bowel disease related to spondyloarthritis has different genetic associations from idiopathic disease and may have a different underlying pathophysiology. Several biomarkers have been shown to reflect response to anti-TNF therapies in spondyloarthritis e.g. MMP3 and VEGF. However, other surrogates of disease, such as bowel permeability, have yet to be examined.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient has a clinical diagnosis with Crohn's disease, as determined by his/her medical history and confirmation of diagnosis by a gastroenterologist
* Patient has either moderate to severely active Crohn's disease as defined by a CDAI score of > 220 and < 450 at Screening or active inflammatory back pain as defined by a BASDAI ≥ 4
* Subject has failed to respond to an adequate course, is intolerant to, or has contraindication to eitherach of the following therapies: Corticosteroids (Prednisone/Budesonide),MTX or Azathioprine/6-mercaptopurine
* Patient is on stable (≥ 1 month) concurrent therapies for Crohn's disease, including 5-aminosalicylates, prednisone (<20 mg/day), budesonide (<9 mg/day), azathioprine, 6-mercaptopurine, methotrexate, and antibiotics
* If female, patient is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or is of childbearing potential and practicing one of the following methods of birth control:condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD),contraceptives (oral or parenteral) for three months (90 days) prior to study drug administration), a vasectomized partner, total abstinence from sexual intercourse
* If patient is female and of childbearing potential, the results of a serum pregnancy test performed at Screening, prior to the first dose of adalimumab, must be negative
* Patient has Crohn's disease for at least 4 months
* Patient has not taken NSAIDs (including OTC) for ≥2 weeks
* Patient has inflammatory back pain according to the Calin or Rudwaleit criteria
* Patient is able and willing to self-administer sc injections or has available a qualified person(s) to administer sc injections
* Patient is able to give written informed consent and to complete the study requirements.

Exclusion criteria

* Patient has current diagnosis of colitis other than Crohn's disease
* Patient has symptomatic known strictures
* Surgical bowel resections within the past 6 months or is planning any resection at any time point while enrolled in the study
* Ostomy or ileoanal pouch
* Short bowel syndrome as determined by the investigator
* Patient has received prior treatment with intravenous immunoglobulin or any investigational agents within four weeks of Baseline, or five half-lives of the product, whichever was longer
* Patient has been previously treated with total lymphoid irradiation or anti-CD4 or CAMPATH 1H monoclonal antibodies resulting in persistent CD4 lymphopenia (CD4 lymphocytes < 500/mm3)
* Patient was previously exposed to a biologic TNF-inhibitor
* Patient has a history of cancer or lymphoproliferative disease other than: Successfully and completely treated Cervical dysplasia, with no recurrence within the last five years
* Has a history of uncontrolled diabetes, unstable ischemic heart disease, congestive heart failure, New York Heart Association (NYHA) III, IV, recent stroke (within three months), chronic leg ulcer and any other condition (e.g., indwelling urinary catheter) which, in the opinion of the Investigator, would put the subject at risk by participation in the protocol or who would make the subject unsuitable for the study
* Positive serology for hepatitis B indicating acute or chronic infection
* Subject is known to have immune deficiency, history of human immunodeficiency virus (HIV) or is immunocompromised
* Persistent or recurrent or severe infections requiring hospitalization or treatment with intra-venous (IV) antibiotics within 30 days, or oral antibiotics within 14 days, prior to Baseline
* Female subjects who are pregnant or breastfeeding
* Has a history of an allergic reaction or significant sensitivity to constituents of adalimumab
* Has a history of clinically significant drug or alcohol abuse in the last year
* Previous diagnosis or signs of central nervous system demyelinating diseases (e.g., optic neuritis, visual disturbance, gait disorder/ataxia, facial paresis, apraxia)
* Patient has a history of active tuberculosis (TB), histoplasmosis or listeriosis, or other currently active infections suggestive of significant or profound immunosuppression, such as Pneumocystis carinii, aspergillosis or other systemic infections
* Patient has latent TB (positive PPD skin test) or has other risk factors for the activation of latent TB, e.g. previous exposure to TB, and has not initiated TB prophylaxis prior to the first adalimumab treatment. In either case, the Principal Investigator (sponsor) must be contacted before initiating the study treatment (see Section 5.6.4, "Screening for Latent Tuberculosis)
* Subjects will be excluded if the CXR is found to have changes suggestive of old healed tuberculous lesion (e.g. calcified nodule, fibrotic scar, apical or basilar pleural thickening etc.)
* Patient has any condition that would prevent participation or completion in this study, including language limitation or possibility that the patient will not be available for the complete study period
* Patient, in the opinion of the principal investigator, is unlikely to comply with the study protocol or is unsuitable for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome measure will be the Ankylosing Spondylitis Assessment Study group 20 (ASAS 20) response at 24 weeks. | 24 weeks

SECONDARY OUTCOMES:
ASAS 20 response | 12 weeks
ASAS 40, 50, 70, 5/6 responses | 12 and 24 weeks
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 12 and 24 weeks
Bath Ankylosing Spondylitis Functional Index (BASFI) | 12 and 24 weeks
Patient Global Assessment of arthritic and CD-related disease activity | 12 and 24 weeks
Total Back Pain | 12 and 24 weeks
Nocturnal Back Pain | 12 and 24 weeks
Erythrocyte sedimentation rate (ESR)/C-reactive protein (CRP) | 12 and 24 weeks
Patient Acceptable Symptom State (PASS) assessments | 12 and 24 weeks
Spinal mobility assessment | 2 and 24 weeks
Enthesitis assessment | 12 and 24 weeks
Crohn's Disease Activity Index (CDAI) | 12 and 24 weeks
Short form 36 (SF-36™) | 12 and 24 weeks
Helplessness scale | 12 and 24 weeks
Spondyloarthritis Research Consortium of Canada Magnetic Resonance Imaging Index (SPARCC MRI) | 24 weeks
Serum biomarkers matrix metalloproteinase 3 (MMP3), vascular endothelial growth factor (VEGF), DKK-1, Wnt, RANKL, OPG and cytokines (e.g. IL17, IL23, IL18) | 12 and 24 weeks
Bowel permeability | 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Walter P Maksymowych, FRCP(C), Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada